CLINICAL TRIAL: NCT05887466
Title: A Single Center, Open, Single Dosing, Dose-escalation, Phase 1/2a Study to Evaluate the Safety and Exploratory Efficacy of Embryonic Stem Cell-derived A9 Dopamine Progenitor Cell (A9-DPC) Therapy in Patients With Parkinson's Disease
Brief Title: Study to Evaluate the Safety and Efficacy of ESC-derived Dopamine Progenitor Cell Therapy in PD Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.Biomedics Co., Ltd. (Industry)
Collaborators: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-PD-001
Record Dates: First submitted 2023-04-09; First posted 2023-06-02 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 3+3 rule-based method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Group (Experimental): 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Study group : 6 subjects
  3. Dosage: 3.15X10^6 cells/body (6 tracks in total, 52.5X10^4 cells per track)
  Interventions: Biological: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) Low Dose
- High Dose Group (Experimental): 1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Study group : 6 subjects
  3. Dosage: 6.30X10^6 cells/body (6 tracks in total, 105X10^4 cells per track)
  Interventions: Biological: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) High Dose

INTERVENTIONS:
Biological: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) Low Dose — Biological/Vaccine: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)_Low Dose
  1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Main ingredients and quantities: A9-DPC -Low Dose :
     7.0X10^6 cells (Use 3.15X10^6 cells of this)
  3. Formulation: milky white cell suspension
  4. Storage method: Refrigerated storage (5±3#)
  5. Expiration date: within 36 hours of manufacture
  6. Frequency: single dosing
  7. Method: The subject pierces a burr hole in the skull on the day of surgery. Then the cells are injected at a predetermined stem cell administration point of the putamen in the brain of the subject. One side is administered in three tracks per putamen (6 tracks total brain). Do the same for the other side.
  Arms: Low Dose Group
Biological: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) High Dose — Biological/Vaccine: Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)_High Dose
  1. IP Name : Allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC)
  2. Main ingredients and quantities: A9-DPC -High Dose :
     1.4X10^7 cells (Use 6.30X10^6 cells of this)
  3. Formulation: milky white cell suspension
  4. Storage method: Refrigerated storage (5±3#)
  5. Expiration date: within 36 hours of manufacture
  6. Frequency: single dosing
  7. Method: The subject pierces a burr hole in the skull on the day of surgery. Then the cells are injected at a predetermined stem cell administration point of the putamen in the brain of the subject. One side is administered in three tracks per putamen (6 tracks total brain). Do the same for the other side.
  Arms: High Dose Group

SUMMARY:
Indication: Patients who were diagnosed with Parkinson's disease ≥ 5 years ago.

Purpose: To find the maximum tolerable dose and evaluate the safety and exploratory efficacy of allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) therapy in patients who were diagnosed with Parkinson's disease ≥ 5 years ago, as a treatment for delaying or stopping the progression of Parkinson's disease or inducing recovery of damaged brain.

Number of Subjects: Up to 12 subjects. [Low dose] 3.15X10^6 cells/body: 6 subjects. [High dose] 6.30X10^6 cells/body: 6 subjects.

Study Design: Single center, open, single dosing, dose-escalation, phase 1/2a study

Endpoints:

[Primary Safety Endpoints]

1. Occurrence of treatment-emergent adverse events (TEAEs) after administration of the IP
2. Failure or rejection of transplantation and occurrence of bleeding and infection at Week 12 (3months), Week 24 (6months), Week 48 (12months) and Week 96 (24months) after administration of the IP
3. Occurrence of adverse event of special interest (AESI)* after administration of the IP

   * AESI: a) death, b) generation of a neoplasm or malignant tumor in tissues or organs, c) onset of an immune reaction including worsening of a previous autoimmune disease or new occurrence, and d) other delayed adverse events related to this embryonic stem cell treatment.

DETAILED DESCRIPTION:
Study Period: Approximately 35 months from the date of approval by the Institutional Review Board (IRB) (However, it can be extended depending on the subject enrollment period or the time to study closure)

Indication: Patients who were diagnosed with Parkinson's disease ≥ 5 years ago

Purpose: To find the maximum tolerable dose and evaluate the safety and exploratory efficacy of allogenic embryonic stem cell-derived A9 dopamine progenitor cell (A9-DPC) therapy in patients who were diagnosed with Parkinson's disease ≥ 5 years ago, as a treatment for delaying or stopping the progression of Parkinson's disease or inducing recovery of damaged brain.

Number of Subjects: Up to 12 subjects [Low dose] Dose: 3.15X10^6 cells/body Study group(A9-DPC): 6 subjects [High dose] Dose: 6.30X10^6 cells/body Study group(A9-DPC): 6 subjects

Study Design: Single center, open, single dosing, dose-escalation, phase 1/2a study

Endpoints:

[Primary Safety Endpoints]

1. Occurrence of treatment-emergent adverse events (TEAEs) after administration of the IP
2. Failure or rejection of transplantation and occurrence of bleeding and infection at Week 12 (3 months), Week 24 (6 months), Week 48 (12 months) and Week 96 (24 months) after administration of the IP
3. Occurrence of adverse event of special interest (AESI)* after administration of the IP *AESI: a) death, b) generation of a neoplasm or malignant tumor in tissues or organs, c) onset of an immune reaction including worsening of a previous autoimmune disease or new occurrence, and d) other delayed adverse events related to this embryonic stem cell treatment.

[Exploratory Efficacy Endpoints]

1. Change in the following clinical endpoints at Week 4 (1 month), Week 12 (3 months), Week 24 (6 months), Week 36 (9 months), Week 48 (12 months), Week 72 (18 months) and Week 96 (24 months) after administration of the IP compared to screening

1. MDS-UPDRS Total Score, part Ⅲ & part Ⅳ (defined on/off)
2. K-MMSE
3. Seoul Neuropsychological screening battery (SNSB, Screening & Week 96 (24 months))
4. Hoehn & Yahr scale

2. Change in the following clinical endpoints at Week 4 (1 month), Week 12 (3 months), Week 24 (6 months), Week 36 (9 months), Week 48 (12 months), Week 72 (18 months) and Week 96 (24 months) after administration of the IP compared to baseline

1. K-MoCA
2. Parkinson's Questionnaire (PDQ-39)
3. Schwab and England ADL scale (SEADL) 4Non-Motor Symptoms Scale for Parkinson's Disease (NMS)

3. Change in Graft size through MRI at Week 12 (3 months), Week 24 (6 months), Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to baseline 4. Change in Cerebral FDG uptake and Striatal FDG uptake at Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to baseline 5. Change in density of dopamine transporters as measured by FP-CIT PET at Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to screening 6. Percentage of subjects who used concomitant medication related to Parkinson-mobility or Parkinson-Non-mobility during the whole clinical trial period and change in dose of each concomitant medication (per component) at 12 week intervals compared to the dose of each concomitant medication (per component) from the date of administration of IP to Week 12.

7. Changes in the following clinical evaluation variables confirmed through the Parkinson's Disease diary at 48 weeks (12 months), 72 weeks (18 months), and 96 weeks (24 months) after administration of the investigational drug compared to baseline:

1. Total waking time
2. Total on-time
3. Total off-time
4. Total dyskinesia time

[Other Safety Endpoints]

1. Vital signs
2. Laboratory tests
3. Physical examination

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease based on UK PD Society Brain Bank criteria at the time of the screening visit
* Patient with Parkinson's disease at the age of 50 to 75 years old at the time of the screening visit
* Patient who was diagnosed with Parkinson' disease ≥ 5 years ago at the time of the screening visit
* Patient on a stable dose of medicine such as levodopa for ≥ 3 months before screening who has wearing off for ≥ 2 hours a day or freezing of gait responding to dopamine supplement or motor complications such as dyskinesia
* At least moderate impairment in activity of daily living (MDS-UPDRS part II ≥13)
* Patient on a stabile dose of standard treatment for Parkinson's disease (e.g., levodopa, dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics, etc.) for ≥ 3 months before screening
* ≥ 40% in L-dopa responsiveness at the time of the screening visit
* Hoehn & Yahr stage ≥ 3 during the off state and stage ≤ 3 during the on state at the time of the screening visit
* Decreased dopamine transporters as measured by FP-CIT PET at the time of the screening visit
* Able to undergo MRI
* Signed consent after being sufficiently informed of the study

Exclusion Criteria:

* Parkinson's disease dementia based on the Movement Disorders Society Task Force criteria
* Parkinsonism plus syndrome confirmed by PET and MRI images at the screening visit
* Patient that does not meet the criteria for Parkinson's disease dementia but has major visual hallucination
* Freezing of gait with no or ambiguous response to L-dopa
* Drug-induced parkinsonism
* History of uncontrolled seizure disorders within 24 weeks before screening
* Congenital developmental delay
* Past or current coagulation factor related diseases at the time of the screening visit
* Ongoing malignancies at the time of the screening visit or diagnosis of malignancies within the past 5 years
* Active tuberculosis, autoimmune disease, or decreased immunity at the time of the screening visit (treatment with chemotherapy within the past 3 years or white blood cell [WBC] <3X10^3 cells/µL)
* Patient diagnosed with diabetes mellitus
* Participation in another clinical trial within 4 weeks before screening
* History of treatment with cell therapy, except for blood transfusion, before study participation
* Side effects to anesthetics, contrast agents, etc.
* Past or current clinically significant diseases in the liver (including liver transplant), kidney, respiratory system, cardiovascular system, etc. or clinically significant laboratory test results at the time of the screening visit

  1. Platelet count < 5.0X10^4/microL
  2. Serum creatinine > 1.5 mg/dL
  3. eGFR < 60 mL/min/1.73 m^2
  4. AST or ALT ≥ 3 x ULN (Upper Limit of Normal)
  5. Total bilirubin ≥ 1.5 x ULN (Upper Limit of Normal)
  6. Hepatitis B or C
  7. Human immunodeficiency virus (HIV) positive
* History of brain surgery
* Pregnant and lactating woman
* Positive pregnancy test at the time of screening; or woman of childbearing potential and man who plan a pregnancy during the study or who do not agree to use clinically appropriate methods of contraception* described below Hormone contraceptives (subdermal contraceptive implants, injections, oral contraceptives, etc.), intrauterine device (IUD) (or intra uterine system [IUS]), subject's or partner's surgical sterilization (vasectomy, tubal ligation, etc.), double barrier method (combined use of barrier methods such as cervical cap or diaphragm in combination with male condom)
* Ineligible for other reasons based on the judgment of the investigator

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) after administration of the IP | Up to 96 Weeks (24 months) after IP administration
  Present frequency and percentage by each dose group about occurrence of treatment-emergent adverse events (TEAEs) after administration of the IP
Failure or rejection of transplantation | Week 12 (3 months)
  Present frequency and percentage by each dose group about failure or rejection of transplantation at Week 12 (3 months) after administration of the IP
Failure or rejection of transplantation | Week 24 (6 months)
  Present frequency and percentage by each dose group about failure or rejection of transplantation at Week 24 (6 months) after administration of the IP
Failure or rejection of transplantation | Week 48 (12 months)
  Present frequency and percentage by each dose group about failure or rejection of transplantation at Week 48 (12 months) after administration of the IP
Failure or rejection of transplantation | Week 96 (24 months)
  Present frequency and percentage by each dose group about failure or rejection of transplantation at Week 96 (24 months) after administration of the IP
Occurrence of bleeding | Week 12 (3 months)
  Present frequency and percentage by each dose group about occurrence of bleeding at Week 12 (3 months) after administration of the IP
Occurrence of bleeding | Week 24 (6 months)
  Present frequency and percentage by each dose group about occurrence of bleeding at Week 24 (6 months) after administration of the IP
Occurrence of bleeding | Week 48 (12 months)
  Present frequency and percentage by each dose group about occurrence of bleeding at Week 48 (12 months) after administration of the IP
Occurrence of bleeding | Week 96 (24 months)
  Present frequency and percentage by each dose group about occurrence of bleeding at Week 96 (24 months) after administration of the IP
Occurrence of infection | Week 12 (3 months)
  Present frequency and percentage by each dose group about occurrence of infection at Week 12 (3 months) after administration of the IP
Occurrence of infection | Week 24 (6 months)
  Present frequency and percentage by each dose group about occurrence of infection at Week 24 (6 months) after administration of the IP
Occurrence of infection | Week 48 (12 months)
  Present frequency and percentage by each dose group about occurrence of infection at Week 48 (12 months) after administration of the IP
Occurrence of infection | Week 96 (24 months)
  Present frequency and percentage by each dose group about occurrence of infection at Week 96 (24 months) after administration of the IP
Occurrence of adverse event of special interest (AESI)* after administration of the IP | Up to 96 Weeks (24 months) after IP administration
  Present frequency and percentage by each dose group about occurrence of adverse event of special interest (AESI)* after administration of the IP
  *AESI: a) death, b) generation of a neoplasm or malignant tumor in tissues or organs, c) onset of an immune reaction including worsening of a previous autoimmune disease or new occurrence, and d) other delayed adverse events related to this embryonic stem cell treatment.

SECONDARY OUTCOMES:
Change in the MDS-UPDRS Total Score, part Ⅲ (defined on/off) & part Ⅳ | -Day 14 to -Day 4, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the MDS-UPDRS Total Scores, part Ⅲ (defined on/off) & part Ⅳ up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 14 to -Day 4).
  * Defined-on condition: condition that the most positive functional effect, as agreed by the subject and the tester, after treatment with drugs for controlling the symptoms of Parkinson's disease
  * Defined-off condition: condition after 12 hours off drugs for controlling the symptoms of Parkinson's disease
Change in the K-MMSE | -Day 14 to -Day 4, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the K-MMSE up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 14 to -Day 4).
Change in the Seoul Neuropsychological screening battery (SNSB, Screening & Week 96 (24 months)) | -Day 14 to -Day 4, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the Seoul Neuropsychological Screening battery (SNSB) between baseline (-Day 14 to -Day 4) and 96 Weeks (24 months) after IP administration.
Hoehn & Yahr scale | Day 14 to -Day 4, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Change in the Hoehn & Yahr scale
Change in the K-MoCA | -Day 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the K-MoCA up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 2).
Change in the Parkinson's Questionnaire (PDQ-39) | -Day 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the Parkinson's Questionnaire (PDQ-39) up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 2).
Change in the Schwab and England ADL scale (SEADL) | -Day 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the Schwab and England ADL scale (SEADL) up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 2).
Change in the Non-Motor Symptoms Scale for Parkinson's Disease (NMS) | -Day 2, Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about changes in the Non-Motor Symptoms Scale for Parkinson's Disease (NMS) up to 96 Weeks (24 months) after IP administration compared to baseline (-Day 2).
Change in Graft size through MRI | -Day 2, Week 12, Week 24, Week 48, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about change in Graft size through MRI at Week 12 (3 months), Week 24 (6 months), Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to baseline (-Day 2)
Change in Cerebral FDG uptake and Striatal FDG uptake | -Day 2, Week 48, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about change in Cerebral FDG uptake and Striatal FDG uptake at Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to baseline (-Day 2)
Change in density of dopamine transporters as measured by FP-CIT PET | -Day 14 to -Day 4, Week 48, Week 96
  Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about change in density of dopamine transporters as measured by FP-CIT PET at Week 48 (12 months) and Week 96 (24 months) after administration of the IP compared to screening (-Day 14 to -Day 4)
Percentage of subjects who used concomitant medication related to Parkinson-mobility or Parkinson-Non-mobility during the whole clinical trial period and Change in dose of each concomitant medication (per component) | Day 0 (Postoperative day #0), Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present the frequency and percentage use of concomitant medication related to Parkinson-mobility or Parkinson-Non-mobility during the whole clinical trial period by each dose group.
  Also Present descriptive statistics (number of subjects, average, standard deviation, median, minimum, maximum) by each dose group about change in dose of each concomitant medication (per component) at 12 week intervals compared to the dose of each concomitant medication (per component) from the date of administration of IP to Week 12.
Parkinson's Disease diary | Day 0 (POD #0), Week 48, Week 72, Week 96
  Changes in the following clinical evaluation variables confirmed through the Parkinson's Disease diary at 48 weeks (12 months), 72 weeks (18 months), and 96 weeks (24 months) after administration of the investigational drug compared to baseline: 1) Total waking time: total waking hours [hours], 2) Total on-time: hours with drug effect [hours], 3)Total off-time: hours without drug effect [hours], 4)Total dyskinesia time: hours with dyskinesia [hours]

OTHER OUTCOMES:
Vital signs | -Day14 to -Day 4, -Day 2, Day 0 (Postoperative day #0), Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistcs(number of subjects, average, standard deviation, median, minimum, maximum) by each dose group for each point in time
Laboratory tests | -Day 14 to -Day 4, Day 0 (Postoperative day #0), Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistcs(number of subjects, average, standard deviation, median, minimum, maximum) by each dose group for each point in time
Physical examination | -Day 14 to -Day 4, -Day 2, Day 0 (Post operative day #0), Week 4, Week 12, Week 24, Week 36, Week 48, Week 72, Week 96
  Present descriptive statistcs(number of subjects, average, standard deviation, median, minimum, maximum) by each dose group for each point in time

CONTACTS AND LOCATIONS:
Overall Officials: Phil-hyu Lee, MD, Ph.D, Principal Investigator — Yonsei Universitiy Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowland NC, Starr PA, Larson PS, Ostrem JL, Marks WJ Jr, Lim DA. Combining cell transplants or gene therapy with deep brain stimulation for Parkinson's disease. Mov Disord. 2015 Feb;30(2):190-5. doi: 10.1002/mds.26083. Epub 2014 Dec 17. PMID 25521796
- [Background] Schweitzer JS, Song B, Herrington TM, Park TY, Lee N, Ko S, Jeon J, Cha Y, Kim K, Li Q, Henchcliffe C, Kaplitt M, Neff C, Rapalino O, Seo H, Lee IH, Kim J, Kim T, Petsko GA, Ritz J, Cohen BM, Kong SW, Leblanc P, Carter BS, Kim KS. Personalized iPSC-Derived Dopamine Progenitor Cells for Parkinson's Disease. N Engl J Med. 2020 May 14;382(20):1926-1932. doi: 10.1056/NEJMoa1915872. PMID 32402162
- [Background] Barker RA, Drouin-Ouellet J, Parmar M. Cell-based therapies for Parkinson disease-past insights and future potential. Nat Rev Neurol. 2015 Sep;11(9):492-503. doi: 10.1038/nrneurol.2015.123. Epub 2015 Aug 4. PMID 26240036
- [Background] Kikuchi T, Morizane A, Doi D, Magotani H, Onoe H, Hayashi T, Mizuma H, Takara S, Takahashi R, Inoue H, Morita S, Yamamoto M, Okita K, Nakagawa M, Parmar M, Takahashi J. Human iPS cell-derived dopaminergic neurons function in a primate Parkinson's disease model. Nature. 2017 Aug 30;548(7669):592-596. doi: 10.1038/nature23664. PMID 28858313
- [Background] Mendez I, Sanchez-Pernaute R, Cooper O, Vinuela A, Ferrari D, Bjorklund L, Dagher A, Isacson O. Cell type analysis of functional fetal dopamine cell suspension transplants in the striatum and substantia nigra of patients with Parkinson's disease. Brain. 2005 Jul;128(Pt 7):1498-510. doi: 10.1093/brain/awh510. Epub 2005 May 4. PMID 15872020
- [Background] Parmar M, Grealish S, Henchcliffe C. The future of stem cell therapies for Parkinson disease. Nat Rev Neurosci. 2020 Feb;21(2):103-115. doi: 10.1038/s41583-019-0257-7. Epub 2020 Jan 6. PMID 31907406
- [Background] Barker RA; TRANSEURO consortium. Designing stem-cell-based dopamine cell replacement trials for Parkinson's disease. Nat Med. 2019 Jul;25(7):1045-1053. doi: 10.1038/s41591-019-0507-2. Epub 2019 Jul 1. PMID 31263283
- [Background] Dubois B, Burn D, Goetz C, Aarsland D, Brown RG, Broe GA, Dickson D, Duyckaerts C, Cummings J, Gauthier S, Korczyn A, Lees A, Levy R, Litvan I, Mizuno Y, McKeith IG, Olanow CW, Poewe W, Sampaio C, Tolosa E, Emre M. Diagnostic procedures for Parkinson's disease dementia: recommendations from the movement disorder society task force. Mov Disord. 2007 Dec;22(16):2314-24. doi: 10.1002/mds.21844. PMID 18098298
- [Background] Baek MJ, Kim K, Park YH, Kim S. The Validity and Reliability of the Mini-Mental State Examination-2 for Detecting Mild Cognitive Impairment and Alzheimer's Disease in a Korean Population. PLoS One. 2016 Sep 26;11(9):e0163792. doi: 10.1371/journal.pone.0163792. eCollection 2016. PMID 27668883
- [Background] Goetz CG, Poewe W, Rascol O, Sampaio C, Stebbins GT, Counsell C, Giladi N, Holloway RG, Moore CG, Wenning GK, Yahr MD, Seidl L; Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. Movement Disorder Society Task Force report on the Hoehn and Yahr staging scale: status and recommendations. Mov Disord. 2004 Sep;19(9):1020-8. doi: 10.1002/mds.20213. PMID 15372591
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression, and mortality. 1967. Neurology. 2001 Nov;57(10 Suppl 3):S11-26. No abstract available. PMID 11775596
- [Background] Koh SB, Kim JW, Ma HI, Ahn TB, Cho JW, Lee PH, Chung SJ, Kim JS, Kwon DY, Baik JS. Validation of the korean-version of the nonmotor symptoms scale for Parkinson's disease. J Clin Neurol. 2012 Dec;8(4):276-83. doi: 10.3988/jcn.2012.8.4.276. Epub 2012 Dec 21. PMID 23323136
- [Background] Shulman LM, Armstrong M, Ellis T, Gruber-Baldini A, Horak F, Nieuwboer A, Parashos S, Post B, Rogers M, Siderowf A, Goetz CG, Schrag A, Stebbins GT, Martinez-Martin P. Disability Rating Scales in Parkinson's Disease: Critique and Recommendations. Mov Disord. 2016 Oct;31(10):1455-1465. doi: 10.1002/mds.26649. PMID 27193358
- [Background] Park HJ, Sohng KY, Kim S. Validation of the Korean version of the 39-Item Parkinson's Disease Questionnaire (PDQ-39). Asian Nurs Res (Korean Soc Nurs Sci). 2014 Mar;8(1):67-74. doi: 10.1016/j.anr.2014.02.004. Epub 2014 Mar 6. PMID 25030495
- [Background] Kefalopoulou Z, Politis M, Piccini P, Mencacci N, Bhatia K, Jahanshahi M, Widner H, Rehncrona S, Brundin P, Bjorklund A, Lindvall O, Limousin P, Quinn N, Foltynie T. Long-term clinical outcome of fetal cell transplantation for Parkinson disease: two case reports. JAMA Neurol. 2014 Jan;71(1):83-7. doi: 10.1001/jamaneurol.2013.4749. PMID 24217017
- [Background] Rasiah NP, Maheshwary R, Kwon CS, Bloomstein JD, Girgis F. Complications of Deep Brain Stimulation for Parkinson Disease and Relationship between Micro-electrode tracks and hemorrhage: Systematic Review and Meta-Analysis. World Neurosurg. 2023 Mar;171:e8-e23. doi: 10.1016/j.wneu.2022.10.034. Epub 2022 Oct 13. PMID 36244666
- [Background] Li W, Englund E, Widner H, Mattsson B, van Westen D, Latt J, Rehncrona S, Brundin P, Bjorklund A, Lindvall O, Li JY. Extensive graft-derived dopaminergic innervation is maintained 24 years after transplantation in the degenerating parkinsonian brain. Proc Natl Acad Sci U S A. 2016 Jun 7;113(23):6544-9. doi: 10.1073/pnas.1605245113. Epub 2016 May 2. PMID 27140603
- [Background] Yasuhara T, Kameda M, Sasaki T, Tajiri N, Date I. Cell Therapy for Parkinson's Disease. Cell Transplant. 2017 Sep;26(9):1551-1559. doi: 10.1177/0963689717735411. PMID 29113472
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Okun MS. Deep-brain stimulation for Parkinson's disease. N Engl J Med. 2012 Oct 18;367(16):1529-38. doi: 10.1056/NEJMct1208070. No abstract available. PMID 23075179
- See also: Phase 1 Safety and Tolerability Study of MSK-DA01 Cell Therapy for Advanced Parkinson's Disease. — http://clinicaltrials.gov/ct2/show/record/NCT04802733.